CLINICAL TRIAL: NCT02562924
Title: An Open-label, Prospective, Randomized, Pilot Clinical Study to Study the Efficacy of MEDIHONEY® Rinses Compared to Intranasal Corticosteroid Rinses in Chronic Rhinosinusitis With Nasal Polyposis After Functional Endoscopic Sinus Surgery
Brief Title: The Efficacy of MEDIHONEY® for Chronic Rhinosinusitis With Nasal Polyposis After Functional Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Gary Landrigan, MD, Associate Professor of Surgery, Division of Otolaryngology, Department of Surgery, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHRMS 15-010
Record Dates: First submitted 2015-04-21; First posted 2015-09-29 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-09

CONDITIONS: Chronic Sinusitis; Nasal Polyposis
Keywords: MEDIHONEY; Chronic Rhinosinusitis With Nasal Polyposis; Functional Endoscopic Sinus Surgery
MeSH Terms: conditions — Nasal Polyps | interventions — Budesonide; Prednisone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Budesonide rinse group (Active Comparator): 1a. Days 0-7: 40 mg prednisone daily, saline sinus rinse 4 times daily, nasal saline spray q 1 hour while awake b. Days 7-91: 8oz saline/budesonide sinus rinse BID (twice daily) c. After day 91: i. In case endoscopy shows any polyps, edema or discharge: Decrease volume to 4 oz budesonide/saline rinse BID. Continue until day 182 ii. In case endoscopy shows no polyps, edema and discharge: Decrease volume to 4 oz budesonide/saline rinse once daily.
  Reevaluate at day 119:
  1. In case endoscopy shows any polyps, edema or discharge: Return to the initial regimen as per 1.c.i till day 182.
  2. In case endoscopy shows no polyps, edema and discharge: Continue as per 1.c.ii till day 182.
  Interventions: Drug: Budesonide; Drug: Normal saline sinus rinse; Drug: Prednisone; Procedure: Endoscopic sinus surgery; Drug: nasal saline spray
- MEDIHONEY® rinse alone group (Experimental): 1. Days 0-7: Same as 1a;
  2. Days 7-91: 8oz saline sinus rinse followed with 0.5oz of MEDIHONEY® in 50 cc of normal saline.
  3. After day 91:
  i. In case endoscopy shows any polyps, edema or discharge: Decrease volume to 4 oz saline rinse followed with the 50cc of the MEDIHONEY®rinse BID. Continue until day 182 ii. In case endoscopy shows no polyps, edema and discharge: Decrease volume to 4 oz saline rinse followed with the 50cc of the MEDIHONEY®rinse once daily. Reevaluate at day 119:
  1. In case endoscopy shows any polyps, edema or discharge: Return to the initial regimen as per 1.c.i till day 182.
  2. In case endoscopy shows no polyps, edema and discharge: Continue as per 1.c.ii till day 182.
  Interventions: Device: MEDIHONEY®; Drug: Normal saline sinus rinse; Drug: Prednisone; Procedure: Endoscopic sinus surgery; Drug: nasal saline spray
- MEDIHONEY® and budesonide rinse group (Experimental): 1. Days 0-7: Same as 1a.;
  2. Days 7-91: 8oz saline/budesonide sinus rinse followed by 0.5oz of MEDIHONEY® in 50 cc of normal saline BID.
  3. After day 91:
  i. In case endoscopy shows any polyps, edema or discharge: Decrease volume to 4 oz budesonide/saline rinse followed with 50cc of the MEDIHONEY® rinse BID. Continue with this regimen till day 182.
  ii. In case endoscopy shows no polyps, edema and discharge: Decrease volume to 4 oz budesonide/saline rinse followed with 50cc of the MEDIHONEY® rinse once a day.
  Reevaluate at day 119:
  1. In case endoscopy shows any polyps, edema or discharge: Return to the initial regimen as per 3.c.i till day 182.
  2. In case endoscopy shows no polyps, edema and discharge: Continue as per 3.c.ii till day 182.
  Interventions: Device: MEDIHONEY®; Drug: Budesonide; Drug: Normal saline sinus rinse; Drug: Prednisone; Procedure: Endoscopic sinus surgery; Drug: nasal saline spray

INTERVENTIONS:
Device: MEDIHONEY® — MEDIHONEY® is a seminatural product with antibacterial and anti-inflammatory properties
  Arms: MEDIHONEY® and budesonide rinse group; MEDIHONEY® rinse alone group
Drug: Budesonide — Topical steroid
  Arms: Budesonide rinse group; MEDIHONEY® and budesonide rinse group
Drug: Normal saline sinus rinse — 8 oz or 4 oz of normal saline with NeilMed sinus rinse bottle
Drug: Prednisone — Post-operatively, 40 mg daily for 7 days
Procedure: Endoscopic sinus surgery — Endoscopic sinus surgery to debride polyps and establish adequate sinus drainage
Drug: nasal saline spray — saline nasal mist every hour while awake

SUMMARY:
This study will assess the effectiveness of MEDIHONEY® sinus rinses (alone or in combination with intranasal corticosteroids) vs. intranasal corticosteroid sinus rinses on mucosal healing and polyp recurrence in the post-operative period following functional endoscopic sinus surgery.

DETAILED DESCRIPTION:
In patients with refractory CRSwNP, functional endoscopic sinus surgery (FESS), is intended to restore physiologic sinus ventilation and drainage, which can facilitate the gradual resolution of mucosal disease. However, because FESS does not directly treat the underlying inflammatory disorder, a successful sinus surgery must be followed by medical maintenance therapy to control inflammatory processes.

The current mainstay of treatment of CRSwNP includes antibiotics and topical and systemic steroids. There is evidence that administration of systemic steroids in the postoperative period for patients who have polyps may have a significant impact on their postoperative course. However, the chance of significant side effects increases with the dose and duration of treatment and therefore the minimum dose necessary to control the disease should be given. Antibiotics also have their limited but documented side effects and can induce resistance.

A semi-natural product like manuka honey (brand name MEDIHONEY®), with antibacterial and anti-inflammatory properties, might prove as a useful alternative since it has no major adverse events documented in the literature, does not induce resistance and is effective against resistant pathogens common in this patient population.

This study is a prospective, randomized, pilot clinical trial that will determine if the use of MEDIHONEY® sinus rinses (alone or in combination with intranasal steroids) in the postoperative period enhances recovery and prevents polyp recurrence in patients after functional endoscopic sinus surgery (FESS), compared with the standard regimen of topical corticosteroid sinus rinses. The study will collect and compare subjective and objective efficacy assessments of both types of rinses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;

2. Diagnosis of CRSwNP based on the following criteria:

* Pattern of symptoms:

  i. Symptoms present for ≥12 wk
* Symptoms for diagnosis: Requires ≥2 of the following symptoms:

  i. Anterior and/or posterior mucopurulent drainage; ii. Nasal obstruction; iii. Facial pain/pressure/fullness;
* Objective documentation: Requires both:

  1. Endoscopy to verify the presence of polyps in middle meatus and document presence of inflammation, such as discolored mucus or edema of middle meatus or ethmoid area; and
  2. Evidence of rhinosinusitis on imaging by CT (1 obvious polypoid tissue or sinus opacification and/or at least 2mm of mucosal thickening).
* Failed medical management (i.e. refractory CRSwNP) and eligible for FESS.

Exclusion Criteria:

1. Contraindications to oral prednisone or known hypersensitivity to any study medications;
2. Churg Strauss disorder;
3. abnormalities of mucociliary clearance (cystic fibrosis, primary ciliary dyskinesia and Young's syndrome);
4. Diagnosed immunodeficiency;
5. Aspirin-induced asthma (ASA) (aka Samter triad) (a triad of asthma, aspirin and NSAID sensitivity, and nasal/ethmoidal polyposis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary P Landrigan, MD, Principal Investigator — University of Vermont Medical Center
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects were enrolled prior to surgery (day 0). Days 0-7 all subjects were treated with oral prednisone once daily, nasal saline irrigation four times daily, and nasal saline misting hourly while awake. Assignment to each arm occurred on day 7. Three enrolled subjects withdrew prior to assignment because they elected to not undergo surgery.
Groups:
- Budesonide Rinse Group: 1a. Days 0-7: 40 mg prednisone daily, saline sinus rinse 4 times daily, nasal saline spray hourly while awake b. Days 7-91: 8oz saline/budesonide sinus rinse BID c. After day 91: i. In case endoscopy shows any polyps, edema or discharge: Decrease volume to 4 oz budesonide/saline rinse BID. Continue until day 182 ii. In case endoscopy shows no polyps, edema and discharge: Decrease volume to 4 oz budesonide/saline rinse once daily.
  Reevaluate at day 119:
  1. In case endoscopy shows any polyps, edema or discharge: Return to the initial regimen as per 1.c.i till day 182.
  2. In case endoscopy shows no polyps, edema and discharge: Continue as per 1.c.ii till day 182.
  Budesonide: Topical steroid Normal saline sinus rinse: 8 oz or 4 oz normal saline with NeilMed sinus rinse bottle Prednisone: Post-operatively 40 mg daily for 7 days Endoscopic sinus surgery: Surgery to debride polyps and establish adequate sinus drainage Nasal saline spray: saline nasal mist every hour while awake
- MEDIHONEY® Rinse Alone Group: 1. Days 0-7: Same as 1a
  2. Days 7-91: 8oz saline sinus rinse followed with 0.5oz of MEDIHONEY® in 50 cc of normal saline
  3. After day 91:
  i. In case endoscopy shows any polyps, edema or discharge: Decrease volume to 4 oz saline rinse followed with the 50cc of MEDIHONEY® rinse BID. Continue until day 182 ii. In case endoscopy shows no polyps, edema and discharge: Decrease volume to 4 oz saline rinse followed with the 50cc of MEDIHONEY® rinse once daily.
  Reevaluate at day 119:
  1. In case endoscopy shows any polyps, edema or discharge: Return to the initial regimen as per 1.c.i until day 182
  2. In case endoscopy shows no polyps, edema and discharge: Continue as per 1.c.ii till day 182
  MEDIHONEY®: A seminatural product with antibacterial and anti-inflammatory properties
- MEDIHONEY® and Budesonide Rinse Group: 1. Days 0-7: Same as 1a
  2. Days 7-91: 8oz saline/budesonide sinus rinse followed by 0.5oz of MEDIHONEY® in 50 cc of normal saline BID
  3. After day 91:
  i. In case endoscopy shows any polyps, edema or discharge: Decrease volume to 4 oz budesonide/saline rinse followed with 50cc of the MEDIHONEY® rinse BID. Continue with this regimen till day 182.
  ii. In case endoscopy shows no polyps, edema and discharge: Decrease volume to 4 oz budesonide/saline rinse followed with 50cc of the MEDIHONEY® rinse once a day.
  Reevaluate at day 119:
  1. In case endoscopy shows any polyps, edema or discharge: Return to the initial regimen as per 3.c.i till day 182.
  2. In case endoscopy shows no polyps, edema and discharge: Continue as per 3.c.ii till day 182.
Period: Overall Study
Arm/Group | Budesonide Rinse Group | MEDIHONEY® Rinse Alone Group | MEDIHONEY® and Budesonide Rinse Group
Started | 13 | 12 | 12
Completed | 12 | 1 | 8
Not Completed | 1 | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide Rinse Group | MEDIHONEY® Rinse Alone Group | MEDIHONEY® and Budesonide Rinse Group | Total
Number analyzed (Participants) | 13 | 12 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (19) | 51 (14) | 58 (8) | 56 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 7
  Male | 11 | 8 | 11 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 13 | 12 | 12 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 12 | 37
Current Smoker [Count of Participants; unit: Participants] | 2 | 1 | 1 | 4
Former Smoker [Count of Participants; unit: Participants] | 5 | 4 | 4 | 13
History of Asthma [Count of Participants; unit: Participants] | 7 | 6 | 6 | 19
History of Diabetes [Count of Participants; unit: Participants] | 2 | 0 | 0 | 2
History of Environmental Allergies [Count of Participants; unit: Participants] | 8 | 7 | 7 | 22
History of Bronchiectasis [Count of Participants; unit: Participants] | 1 | 1 | 2 | 4
Lund-Mackay Radiographic Score [Mean (Standard Deviation); unit: units on a scale] — Radiographic scoring system based on pre-operative CT scan. Each sinus (anterior ethmoid, posterior ethmoid, maxillary, frontal, sphenoid) on the left and right are given a score of 0, 1 or 2 for no abnormality, partial opacification, and total opacification, respectively. Additionally, the right and left osteomeatal complexes are scored 0 or 2 for non-obstructed or obstructed, respectively. These values are summed, and a score between 0 and 24 is assigned. The higher the score, the worse the baseline disease.
  units on a scale | 15.8 (6.6) | 14.8 (5.6) | 18.3 (5.2) | 15.6 (6.7)
Baseline Surgery Score [Mean (Standard Deviation); unit: units on a scale] — Score on a scale of 0 to 14 to describe the extent of surgery performed. One point is assigned if that procedure is performed. The 7 possible procedures include anterior ethmoidectomy, frontal recess surgery, middle meatal antrostomy, posterior ethmoidectomy, reduction of middle turbinate, sphenoidectomy, uncinectomy. Scores are assigned for the left and right separately (up to 7 points on each side). A higher score indicates that more surgery was performed.
  units on a scale | 12.8 (1.0) | 13.0 (1.0) | 13.5 (0.9) | 13.1 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lund-Kennedy Endoscopic Scores
Description: Characteristics of each sinonasal cavity are assessed endoscopically to provide a score based on polyp disease, mucosal edema/crusting/scarring and nasal secretions. A score is provided for the left and right. The scores are totaled to provide a number between 0 and 20.
  Polyps: 0 = absence of polyp; 1 = polyps in middle meatus only; 2 = polyps beyond middle meatus Edema: 0 = absent; 1 = mild; 2 = severe Discharge: 0 = no discharge; 1 = clear, thin discharge; 2 = thick, purulent discharge Scarring: 0 = absent; 1 = mild; 2 = severe Crusting: 0 = absent; 1 = mild; 2 = severe
  This scoring system has since been the instrument of choice to endoscopically evaluate outcomes of interventions in non-neoplastic sinonasal disease prospectively over time in research and clinical practice. The higher the score, the worse the outcome. Endoscopy scores from the 3 study groups are compared for the average unit change between baseline and day 119.
Time Frame: 119 days
Population: The population analyzed for this outcome is the population of participants for which we had data points at day 119. Please note that this is different than the number of participants that completed the study (Budesonide: 13 enrolled, 11 analyzed; MEDIHONEY: 12 enrolled, 6 analyzed; MEDIHONEY and budesonide: 12 enrolled, 9 analyzed).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Budesonide Rinse Group | MEDIHONEY® Rinse Alone Group | MEDIHONEY® and Budesonide Rinse Group
Number analyzed (Participants) | 11 | 6 | 9
score on a scale | -8.0 (3.1) | -1.5 (4.6) | -6.9 (3.9)

2. Secondary Outcome: Nasal Drainage Cultures
Description: Nasal drainage cultures from the 3 study groups will be compared for the average percent change between a patient's positive intraoperative cultures compared to the patient's cultures at day 35.
Time Frame: 35 days
Population: This secondary objective describes analyzing quantitative changes in microbiology between day of surgery and post-operative day 35. These data were not collected, but rather the qualitative data (which microorganisms were present) were. Therefore we are not able to complete analysis on this secondary objective.
Arm/Group | Budesonide Rinse Group | MEDIHONEY® Rinse Alone Group | MEDIHONEY® and Budesonide Rinse Group
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in Sinonasal Outcome Test (SNOT-22) Questionnaire Score
Description: The SNOT-22 consists of 22 questions; items 1 to 12 represent the physical problems associated with rhinosinusitis, items 13 to 18 represent the functional limitations, and items 20 to 22 represent the emotional consequences. Each question is scored by the patient from 0 (no problem) to 5 (the problem is as bad as it can be). The overall score can theoretically range from 0 to 110, with higher scores reflecting more severe quality of life impairment as subjectively reported by the patient. Overall SNOT-22 scores from the 3 study groups are compared for the average change in score from baseline to day 119.
Time Frame: 119 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Budesonide Rinse Group | MEDIHONEY® Rinse Alone Group | MEDIHONEY® and Budesonide Rinse Group
Number analyzed (Participants) | 11 | 6 | 9
score on a scale | -22.8 (20.2) | -15.3 (27.4) | -25.6 (16.9)

4. Secondary Outcome: Change in SNOT-22 Nasal Symptom Scores
Description: The SNOT-22 consists of 22 questions; items 1 to 12 represent the physical problems associated with rhinosinusitis, items 13 to 18 represent the functional limitations, and items 20 to 22 represent the emotional consequences. Each question is scored by the patient from 0 (no problem) to 5 (the problem is as bad as it can be).
  The first seven questions relate to nasal symptoms. The nasal symptoms score is calculated by summing the scores for these first seven questions. The range is 0 to 35. Higher scores reflect more severe quality of life impairment as subjectively reported by the patient. The nasal symptom scores from the 3 study groups are compared for the average change in score from baseline to day 119.
Time Frame: 119 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Budesonide Rinse Group | MEDIHONEY® Rinse Alone Group | MEDIHONEY® and Budesonide Rinse Group
Number analyzed (Participants) | 11 | 6 | 9
score on a scale | -10.0 (7.0) | -5.3 (15.5) | -11.7 (7.9)

ADVERSE EVENTS:
Time Frame: Adverse event data was recorded in the form of a modified version of the Common Toxicity Criteria for Adverse Events (CTCAE). This was done at each visit from baseline (pre-surgery) to the 6th visit on day 182.
Arm/Group | Budesonide Rinse Group | MEDIHONEY® Rinse Alone Group | MEDIHONEY® and Budesonide Rinse Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 1/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/13 | 2/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide Rinse Group (N=13) | MEDIHONEY® Rinse Alone Group (N=12) | MEDIHONEY® and Budesonide Rinse Group (N=12)
Nasal Pain (General disorders) | 1 | 0 | 0
Blurred Vision (Eye disorders) | 1 | 0 | 0
Mood alteration (anxiety) (Psychiatric disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Limitations of this study include: non-blinded study, high drop-out rate in one study arm, and lack of quantitative data for sinus cultures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT02562924/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT02562924/SAP_001.pdf